CLINICAL TRIAL: NCT06332690
Title: Imaging Biomarkers of Treatment Response to Dexamethasone Implant in Macular Edema Due to Retinal Vascular Diseases - Diabetic Macular Edema and Retinal Vein Occlusion.
Brief Title: OCT and OCT-Angiography Biomarkers of Treatment Response to Dexamethasone Implant in Macular Edema Due to Retinal Vascular Diseases - DME and RVO
Status: Recruiting | Type: Observational
Sponsor: IRCCS Multimedica (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 514.2021
Record Dates: First submitted 2024-03-17; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Macular Edema; Macular Edema Due to Diabetes Mellitus; Retinal Vein Occlusion
Keywords: Diabetic macular edema; macular edema due to retinal vein occlusion; diabetes mellitus; retinal imaging
MeSH Terms: conditions — Retinal Vein Occlusion; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: dexamethasone implant — Intravitreal dexamethasone implant (Dex) slowly releases steroids into the vitreous over a period of up to 6 months. Dex 0.7 mg (Ozurdex™; Allergan, Irvine, CA, USA) has been used to reduce ME in patients with DR and RVO and its efficacy in terms of best corrected visual acuity (BCVA) improvement and central macular thickness (CMT) reduction has been demonstrated in many different studies.

SUMMARY:
The purpose of this pilot study is to evaluate different imaging parameters in patients with previously treatment-naive DME and ME due to RVO before and after treatment with dexamethasone implant, in order to find specific retinal inflammatory and microvascular biomarkers that may be predictive of treatment outcome.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) and retinal vein occlusion (RVO) are complex multifactorial diseases and the leading causes of visual impairment worldwide. The exact mechanisms leading to Macular Edema (ME) in DR and RVO are not fully understood, actual evidence focuses on the role of inflammation as critical contributing factor in ME pathogenesis and several studies described the association between high levels of systemic and local inflammatory molecules and the development of ME. Even if vascular endothelial growth factor (VEGF) is the most studied factor involved in ME pathogenesis in retinal vascular diseases and the main target of available therapeutic strategies, its role cannot explain alone all the events taking place in the onset and progression of these diseases. VEGF selective inhibition is not sufficient to stop the inflammatory cascade in DR and RVO and anti-VEGF therapies are frequently of transient benefit, especially in DME treatment, needing repeated injections over time and suggesting the involvement of other molecular pathways. Intravitreal corticosteroids block the production of inflammatory mediators (including VEGF) and inhibit leukostasis. In particular, dexamethasone has the highest relative clinical efficacy of any corticosteroid applied to ophthalmology practice. Intravitreal dexamethasone implant (Dex) slowly releases steroids into the vitreous over a period of up to 6 months. Dex 0.7 mg (Ozurdex™; Allergan, Irvine, CA, USA) has been used to reduce ME in patients with DR and RVO and its efficacy in terms of best corrected visual acuity (BCVA) improvement and central macular thickness (CMT) reduction has been demonstrated in many different studies. Thanks to the great advances in retinal imaging technologies of the last years, a new concept of non-invasive "imaging biomarker" of retinal inflammation has emerged and has made its way in the study of patients with DR and RVO. Clinical research has consequently developed great interest in finding specific retinal inflammatory parameters in DR and RVO and there is a growing body of scientific evidence on the importance of this topic. Moreover, the evaluation of these inflammatory biomarkers might be helpful in the prediction of treatment response. Nowadays, main proposed imaging biomarkers of inflammation include subfoveal neuroretinal detachment (SND) and hyperreflective retinal spots (HRS), visible on optical coherence tomography (OCT). SND consists in extracellular fluid accumulation between the outer segments of photoreceptors and the retinal pigment epithelium and is present in approximately 15-30% of eyes with DME and in an even greater number of patients with ME secondary to RVO. The presence of SND has been associated with higher levels of local inflammatory molecules, in particular IL-6. HRS are increased in number in patients with diabetes (with or without DR) and RVO; they have specific characteristics and are thought to represent aggregates of activated microglial cells that progressively migrate from the inner to the outer retina, confirming their role as inflammatory biomarkers. The purpose of this pilot study is to evaluate different imaging parameters in patients with previously treatment-naive DME and ME due to RVO before and after treatment with dexamethasone implant, in order to find specific retinal inflammatory and microvascular biomarkers that may be predictive of treatment outcome. The novelty of this study is a detailed evaluation of multimodal imaging modifications in DME and ME due to RVO after treatment with Dex in order to document its anti-inflammatory effect.

ELIGIBILITY:
Inclusion Criteria:

* previously untreated centre-involving DME or ME secondary to RVO with CMT ≥ 300 μm;
* pseudophakic eyes or eyes with a transparent lens or only initial sclerosis of the lens, in order to obtain good quality retinal imaging
* patient agreement to participate in the study.

Exclusion Criteria:

* any retinal disease other than DR or RVO;

  * a positive history of retinal surgery and/or any other macular/retinal treatment (laser, intravitreal injections of anti-VEGF and/or steroids);
  * cataract surgery within 6 months in the study eye;
  * refractive error > +/- 4D;
  * Advanced glaucoma
  * neurodegenerative diseases (e.g. multiple sclerosis, Alzheimer disease, Parkinson disease, etc.)
  * poor quality of OCT and/or OCT-A images due to significant media opacity or poor patient cooperation.
  * Ocular or periocular infections (including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases
  * Non-intact posterior lens capsule
  * Hypersensitivity to any component of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for intravitreal Dexamethasone implantation for diabetic macular edema and retinal vein occlusion.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Modification of inflammatory biomarkers on OCT and perfusion density parameters on OCT-A at 4 months after surgery (Change measure) | pre-surgery and at 4 months after each surgery (if applicable)
  Evaluate different inflammatory and microvascular parameters on imaging exams (OCT-A, OCT, and FAF) in patients with DME and ME secondary to RVO before and after treatment with intravitreal Dexamethasone implant, in order to identify specific predictive (imaging) biomarkers of treatment.
  If a new surgery is required at 4 months, an additional follow-up will be scheduled 4 months after the second surgery

SECONDARY OUTCOMES:
Initial clinical characteristics in patients with a gain in BCVA (Best Corrected Visual Acuity) of ≥ 5, ≥ 10, and ≥ 15 ETDRS (Early Treatment Diabetic Retinopathy Study) letters. | pre-surgery and up to every 2 months
  Evaluate different inflammatory and microvascular parameters on imaging exams (OCT, OCT-A, and FAF) in patients with improvement in BCVA (≥ 5, ≥ 10, and ≥ 15 ETDRS letters) at the final visit; and in patients showing recurrence during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Stela Vujosevic, MD, Principal Investigator — MultiMedica - IRCCS MultiMedica
Locations (1):
- MultiMedica IRCCS Multimedica, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vujosevic S, Simo R. Local and Systemic Inflammatory Biomarkers of Diabetic Retinopathy: An Integrative Approach. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO68-BIO75. doi: 10.1167/iovs.17-21769. PMID 28510630
- [Result] Jenkins AJ, Joglekar MV, Hardikar AA, Keech AC, O'Neal DN, Januszewski AS. Biomarkers in Diabetic Retinopathy. Rev Diabet Stud. 2015 Spring-Summer;12(1-2):159-95. doi: 10.1900/RDS.2015.12.159. Epub 2015 Aug 10. PMID 26676667
- [Result] Vujosevic S, Bini S, Torresin T, Berton M, Midena G, Parrozzani R, Martini F, Pucci P, Daniele AR, Cavarzeran F, Midena E. HYPERREFLECTIVE RETINAL SPOTS IN NORMAL AND DIABETIC EYES: B-Scan and En Face Spectral Domain Optical Coherence Tomography Evaluation. Retina. 2017 Jun;37(6):1092-1103. doi: 10.1097/IAE.0000000000001304. PMID 27668929
- [Result] Vujosevic S, Torresin T, Bini S, Convento E, Pilotto E, Parrozzani R, Midena E. Imaging retinal inflammatory biomarkers after intravitreal steroid and anti-VEGF treatment in diabetic macular oedema. Acta Ophthalmol. 2017 Aug;95(5):464-471. doi: 10.1111/aos.13294. Epub 2016 Oct 24. PMID 27775223
- [Result] McAllister IL, Vijayasekaran S, Zhang D, McLenachan S, Chen FK, Yu DY. Neuronal degeneration and associated alterations in cytokine and protein in an experimental branch retinal venous occlusion model. Exp Eye Res. 2018 Sep;174:133-146. doi: 10.1016/j.exer.2018.05.025. Epub 2018 May 24. PMID 29803555
- [Result] Boyer DS, Yoon YH, Belfort R Jr, Bandello F, Maturi RK, Augustin AJ, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Three-year, randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1904-14. doi: 10.1016/j.ophtha.2014.04.024. Epub 2014 Jun 4. PMID 24907062
- [Result] Callanan DG, Gupta S, Boyer DS, Ciulla TA, Singer MA, Kuppermann BD, Liu CC, Li XY, Hollander DA, Schiffman RM, Whitcup SM; Ozurdex PLACID Study Group. Dexamethasone intravitreal implant in combination with laser photocoagulation for the treatment of diffuse diabetic macular edema. Ophthalmology. 2013 Sep;120(9):1843-51. doi: 10.1016/j.ophtha.2013.02.018. Epub 2013 May 22. PMID 23706947
- [Result] Haller JA, Bandello F, Belfort R Jr, Blumenkranz MS, Gillies M, Heier J, Loewenstein A, Yoon YH, Jiao J, Li XY, Whitcup SM; Ozurdex GENEVA Study Group; Li J. Dexamethasone intravitreal implant in patients with macular edema related to branch or central retinal vein occlusion twelve-month study results. Ophthalmology. 2011 Dec;118(12):2453-60. doi: 10.1016/j.ophtha.2011.05.014. Epub 2011 Jul 20. PMID 21764136
- [Result] Querques L, Querques G, Lattanzio R, Gigante SR, Del Turco C, Corradetti G, Cascavilla ML, Bandello F. Repeated intravitreal dexamethasone implant (Ozurdex(R)) for retinal vein occlusion. Ophthalmologica. 2013;229(1):21-5. doi: 10.1159/000342160. Epub 2012 Sep 19. PMID 23006995
- [Result] Chang-Lin JE, Attar M, Acheampong AA, Robinson MR, Whitcup SM, Kuppermann BD, Welty D. Pharmacokinetics and pharmacodynamics of a sustained-release dexamethasone intravitreal implant. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):80-6. doi: 10.1167/iovs.10-5285. PMID 20702826
- [Result] Otani T, Kishi S, Maruyama Y. Patterns of diabetic macular edema with optical coherence tomography. Am J Ophthalmol. 1999 Jun;127(6):688-93. doi: 10.1016/s0002-9394(99)00033-1. PMID 10372879
- [Result] Gaucher D, Sebah C, Erginay A, Haouchine B, Tadayoni R, Gaudric A, Massin P. Optical coherence tomography features during the evolution of serous retinal detachment in patients with diabetic macular edema. Am J Ophthalmol. 2008 Feb;145(2):289-296. doi: 10.1016/j.ajo.2007.09.029. Epub 2007 Dec 11. PMID 18054885
- [Result] Catier A, Tadayoni R, Paques M, Erginay A, Haouchine B, Gaudric A, Massin P. Characterization of macular edema from various etiologies by optical coherence tomography. Am J Ophthalmol. 2005 Aug;140(2):200-6. doi: 10.1016/j.ajo.2005.02.053. PMID 15992752
- [Result] Ozdemir H, Karacorlu M, Karacorlu S. Serous macular detachment in diabetic cystoid macular oedema. Acta Ophthalmol Scand. 2005 Feb;83(1):63-6. doi: 10.1111/j.1600-0420.2005.00387.x. PMID 15715559
- [Result] Vujosevic S, Bini S, Midena G, Berton M, Pilotto E, Midena E. Hyperreflective intraretinal spots in diabetics without and with nonproliferative diabetic retinopathy: an in vivo study using spectral domain OCT. J Diabetes Res. 2013;2013:491835. doi: 10.1155/2013/491835. Epub 2013 Dec 9. PMID 24386645